CLINICAL TRIAL: NCT03510793
Title: Changes in the Sublingual Microcirculation Following Aortic Surgery Under Balanced or Total Intravenous Anesthesia: a Prospective Observational Study
Brief Title: Microcirculation and Anesthesia in Vascular Surgery
Status: Completed | Type: Observational
Sponsor: Università Politecnica delle Marche (Other)
Responsible Party: Principal Investigator, Abele Donati, MD, Professor, Università Politecnica delle Marche
Other Study IDs: Vasc2018
Record Dates: First submitted 2018-04-24; First posted 2018-04-27 (Actual); Last update posted 2018-05-03 (Actual); Status verified 2018-04

CONDITIONS: Ischemia Reperfusion Injury; Aortic Aneurysm; Anesthesia
Keywords: microcirculation; aortic aneurysm; anesthesia
MeSH Terms: conditions — Reperfusion Injury; Aortic Aneurysm | interventions — Balanced Anesthesia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Balanced anesthesia: Patients receiving balanced anesthesia (desflurane + remifentanil) according to the attending physician's decision
  Interventions: Drug: balanced anesthesia
- Total intravenous anesthesia: Patients receiving total intravenous anesthesia (TIVA) using propofol + remifentanil with target-controlled infusion according to the attending physician's decision.
  Interventions: Drug: Total intravenous anesthesia

INTERVENTIONS:
Drug: balanced anesthesia — patients undergoing open elective abdominal aortic aneurysm repair will receive balanced (desflurane + remifentanil) anaesthesia
  Groups: Balanced anesthesia
Drug: Total intravenous anesthesia — patients undergoing open elective abdominal aortic aneurysm repair will receive total intravenous (propofol + remifentanil with target-controlled infusion) anesthesia
  Groups: Total intravenous anesthesia

SUMMARY:
Ischemia/reperfusion injury following aortic cross-clamping for vascular surgery leads to systemic hemodynamic and microcirculatory perturbances. The use of different anesthetic regimens may have an impact on tissue perfusion. The aim of this study was to explore changes in microvascular perfusion in patients undergoing elective open abdominal aortic aneurysm repair under balanced or total intravenous anesthesia. Prospective observational study on 40 patients scheduled for elective open infrarenal abdominal aortic aneurysm repair, who received balanced (desflurane + remifentanil, n=20) or total intravenous anesthesia (TIVA, propofol + remifentanil using target-controlled infusion, n=20) according to the clinician's decision. A goal-directed hemodynamic management was applied in all patients. Hemodynamics and arterial/venous blood gases were compared before anesthesia induction (baseline) and at end-surgery. Changes in sublingual microvascular flow and density were assessed with incident dark field illumination imaging. Near infrared spectroscopy was applied on the thenar eminence with a vascular occlusion test (VOT) to assess variations in the peripheral muscle tissue oxygenation and microcirculatory reactivity.

DETAILED DESCRIPTION:
Ischemia/reperfusion (I/R) injury is a common problem in patients undergoing aortic clamping for vascular surgery and may lead to systemic inflammation and organ dysfunction. Increased production of pro-inflammatory molecules and oxidative stress induced by I/R are responsible for microvascular alterations similar to those observed during sepsis, which result in tissue hypoxia. Anesthetics can affect the microcirculation. Propofol causes vasodilation stimulating NO production and decreases microvascular density. A final arteriolar vasodilation could involve a greater oxygen delivery and better perfusion, but a massive dose-dependent vasodilation could lead to a shunt of blood flow with reduced oxygen availability. Volatile anesthetics cause dose-dependent vasodilation too and desflurane, unlike isoflurane and alothane, maintains myocardial, hepatic, intestinal and muscle blood flow. This prospective observational study aims to evaluate the effects of intravenous and balanced anesthesia on sublingual and peripheral muscle microcirculation in patients undergoing elective open abdominal aortic aneurysm repair. This study was approved by the investigator's local ethical committee of Azienda Ospedaliera Universitaria "Ospedali Riuniti" of Ancona, Italy. A written informed consent was obtained from all patients. Patients were eligible if they were scheduled for elective infrarenal abdominal aortic open repair with or without prosthetic aorto-aortic or aorto-bisiliac bypass under general anesthesia. Patients received balanced (desflurane + remifentanil) or total intravenous (TIVA, propofol + remifentanil, with target-controlled infusion) anesthesia according to the attending physician's decision, resulting in two study groups. Spectral entropy was used in monitoring anesthetic depth. A goal-directed hemodynamic management was applied in all patients. Hemodynamics was evaluated with Flotrac/Vigileo (Edwards Lifesciences) monitor according to routine clinical practice. Arterial and central venous blood gases were measured according to routine clinical practice. All measurements were collected before anesthesia induction (baseline) and at end-surgery. Changes in sublingual microvascular flow and density were assessed with incident dark field illumination imaging (Cytocam, Braedius, Amsterdam, NL). After gentle removal of saliva and other secretions with a gauze, the probe was applied to the sublingual region, avoiding excessive pressure. Three sequences of 10 seconds each were recorded in 3 different mucosal areas. Subsequently, clips were analysed offline by AVA software (Automated Vascular Analysis v3.0). The following parameters were calculated for small vessels: microvascular flow index, total vessel density, perfused vessel density, percentage of perfused vessels, flow heterogeneity index. Near infrared spectroscopy (InSpectra, Hutchinson Technology, MN, USA) was applied on the thenar eminence with a vascular occlusion test (VOT) to assess variations in the peripheral muscle tissue oxygenation and microcirculatory reactivity. A probe was applied on the thenar eminence, and, after a 3-minute period of stabilization, tissue O2 saturation (StO2) and tissue haemoglobin index (THI) were recorded. Then arterial inflow was arrested by inflating a sphygmomanometer cuff to 50mmHg above the systolic arterial pressure; the cuff was kept inflated until StO2 decreased to 40% and finally was released. StO2 modifications were continuously recorded during the reperfusion phase until stabilization. The following parameters were extrapolated: StO2 downslope, StO2 upslope, area of hyperemia. Statistics: normality of distribution will be assessed with Kolmogorov-Smirnov test. Data will be expressed as mean±standard deviation or median [1st-3rd quartile], as appropriate. Two-way ANOVA with Sidack's multiple comparisons test or Wilcoxon and Mann-Whitney U test were used to compare variables between the two time points into the same group and between two groups at time-matched points as appropriate. A p value <0.05 was used to indicate statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* elective infrarenal abdominal aortic open repair
* protocol of intraoperative goal-directed therapy
* ASA class I-II-III

Exclusion Criteria:

* age of less than 18 years
* pregnancy
* Endovascular Aneurysm Repair (EVAR)
* concomitant infections
* trauma
* emergency surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult (>18 years old) patients scheduled for elective open aortic aneurysm repair under general anesthesia, who will receive balanced or total intravenous anesthesia according to the attending physician's decision
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2013-09-01 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
change in the microvascular flow index | from baseline (before induction of anesthesia) to end-surgery (before anesthesia suspension)
  Variation in the microvascular flow index, which is a parameter of capillary blood flow quality, calculated for small (diameter <20 microns) vessels in the sublingual microcirculation

SECONDARY OUTCOMES:
change in microvascular density | from baseline (before induction of anesthesia) to end-surgery (before anesthesia suspension)
  Variation in parameters of sublingual total and perfused vessel densities
change in tissue oxygenation | from baseline (before induction of anesthesia) to end-surgery (before anesthesia suspension)
  Variation in skeletal muscle (thenar eminence) StO2
change in microvascular reactivity | from baseline (before induction of anesthesia) to end-surgery (before anesthesia suspension)
  Variation in skeletal muscle (thenar eminence) StO2 upslope, which is the slope of the reperfusion phase during the vascular occlusion test

CONTACTS AND LOCATIONS:
Overall Officials: Abele Donati, Principal Investigator — Università Politecnica delle Marche

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Petros AJ, Bogle RG, Pearson JD. Propofol stimulates nitric oxide release from cultured porcine aortic endothelial cells. Br J Pharmacol. 1993 May;109(1):6-7. doi: 10.1111/j.1476-5381.1993.tb13523.x. PMID 8388302
- [Result] Koch M, De Backer D, Vincent JL, Barvais L, Hennart D, Schmartz D. Effects of propofol on human microcirculation. Br J Anaesth. 2008 Oct;101(4):473-8. doi: 10.1093/bja/aen210. Epub 2008 Jul 23. PMID 18653494
- [Result] O'Riordan J, O'Beirne HA, Young Y, Bellamy MC. Effects of desflurane and isoflurane on splanchnic microcirculation during major surgery. Br J Anaesth. 1997 Jan;78(1):95-6. doi: 10.1093/bja/78.1.95. PMID 9059215
- [Derived] Loggi S, Mininno N, Damiani E, Marini B, Adrario E, Scorcella C, Domizi R, Carsetti A, Pantanetti S, Pagliariccio G, Carbonari L, Donati A. Changes in the sublingual microcirculation following aortic surgery under balanced or total intravenous anaesthesia: a prospective observational study. BMC Anesthesiol. 2019 Jan 5;19(1):1. doi: 10.1186/s12871-018-0673-7. PMID 30611197